CLINICAL TRIAL: NCT04811807
Title: Multicentre Observational Study of Impulsive Behaviours Following Deep Brain Stimulation in Parkinson's Disease
Brief Title: Clinical Response of Impulsivity After Brain Stimulation in Parkinson's Disease
Acronym: CRIPS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other); NHS Greater Glasgow and Clyde (Other); King's College Hospital NHS Trust (Other); Walton Centre NHS Foundation Trust (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other); Oxford University Hospitals NHS Trust (Other); Barking, Havering and Redbridge University Hospitals NHS Trust (Other); Northern Care Alliance NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 285162
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-03

CONDITIONS: Impulsive Behavior; Impulse Disorders; Gambling, Pathological; Eating, Binge; Hoarding Disorder; Hypersexuality; Compulsive Shopping; Dopamine Dysregulation Syndrome; Caregiver Burnout; Parkinson Disease
Keywords: Deep brain stimulation; Parkinson's disease; Impulse control disorders; Impulse control behaviours; compulsive shopping; hypersexuality; binge eating; gambling; walkabouts; hobbyism; Hoarding; punding
MeSH Terms: conditions — Impulsive Behavior; Gambling; Bulimia; Hoarding Disorder; Compulsive Sexual Behavior Disorder; Caregiver Burden; Parkinson Disease; Disruptive, Impulse Control, and Conduct Disorders; Hoarding | interventions — Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Subthalamic Nucleaus Deep brain stimulation — In deep brain stimulation (DBS) therapy, a specific anatomical target in the brain is stimulated via surgically fixed electrodes. These electrodes release electrical currents of a specific voltage, wavelength, and frequency. They are connected via subcutaneous wires to a device called an implantable pulse generator (IPG) which is surgically fixed on chest wall, beneath the clavicle. After electrodes and IPG are successfully installed, a clinician will be able to adjust and modulate the stimulation via a remote device connected to the IPG to obtain a maximum potential benefit. Deep brain stimulation has been used in clinics to treat various neurologic diseases including neurodegenerative disorders, mainly movement disorders.
  Other Names: DBS; Brain stimulation

SUMMARY:
The objective of this prospective observational cohort study is to answer the following clinically important questions:

1. In patients with a pre-operative history of ICBs, what is the likelihood of improvement or deterioration in ICBs post-operatively?
2. What is the risk of developing post-operative de novo ICBs after Subthalamic Nucleus DBS (STN DBS)?
3. Which factors are important in predicting changes in ICBs after STN DBS?
4. What is the impact of ICBs on carer's quality of life QoL and burden?

DETAILED DESCRIPTION:
The study will record outcomes related to ICBs for PD patients who have already been selected for DBS therapy as a routine clinical treatment in participating in DBS operating centre

It is routine practice to assess ICBs before DBS decisions are made, but the manner varies across DBS operating centres. The only additional factor to the routine DBS clinical pathway in this study is that the centres involved will perform assessments in a uniform manner to allow data to be combined. A unified set of clinical assessment scales for Impulsive Control Disorders ICDs and ICBs, as well as other relevant neuropsychiatric symptom assessment, will be added to routine pre- and post-operational clinical assessments for participants.

The primary endpoint of the study is the change in severity of ICBs. If subjects score above 1 in any of given questions on QUIP-RS, or if subjects had disagreement with carers regarding scores, The Parkinson's Impulse-Control Scale, PICs will be triggered. PICs then will be administered by our trained research fellow (AA), over phone or in the clinic.

Other scales to be administered are listed below:

1. Neuropsychiatric Inventory (NPI)
2. General anxiety disorder-7 (GAD-7)
3. Patient Health Questionnaire-9 (PHQ9)
4. Parkinson's disease questionnaire-39 (PDQ-39)
5. EuroQol 5 Dimension (EQ-5D)
6. Clinical Global Impression - Severity scale (CGI-S) at baseline and Clinician's Global Impression - Improvement scale (GGI-I) post-operatively.
7. Zarit Caregiver Burden Scale
8. Work and Social Adjustment Scale
9. UPPS-P Impulsive Behaviour Scale

Assessments will be performed at baseline, 3, 6 and 12 months post-operatively.

Results will be analysed to ascertain potential predictive measures for ICBS development/change.

ELIGIBILITY:
Inclusion Criteria:

* Selected for DBS to treat motor symptoms of Parkinson's disease
* English language fluency

Exclusion Criteria:

* nil

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All potential participants will have been selected by their clinicians for DBS to treat their motor symptoms as routine clinical care. They will be approached during their hospital appointment by their clinical care team, who will be the research link to this study, principal investigator
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
change in severity of ICBs and development of new ICBs | 12 months
Descriptive analysis of recurrence of ICBs in those with history of ICBs using scores on QUIP-RS/PICs | 12 months
Descriptive analysis of de novo cases of Impulsive control disorders ICD/ICBs | 12 months

SECONDARY OUTCOMES:
predictive factors for de novo, recurrence and change in severity of ICD/ICBs | 12 months
change in ICB relate to quality of life in patients and carers | 12 months
change in ICD relates to changes in mood | 12 months
change in ICD relates to change in personality traits | 12 months

IPD SHARING:
Plan to Share IPD: No